CLINICAL TRIAL: NCT03939520
Title: Pragmatic Management of Progressive Disease in Idiopathic Pulmonary Fibrosis: a Randomized Trial
Brief Title: Management of Progressive Disease in Idiopathic Pulmonary Fibrosis
Acronym: PROGRESSION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0029; 2024-511427-34-00 (EU CTIS Number); 2019-004326-19 (EudraCT Number)
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Progressive Idiopathic Pulmonary Fibrosis
Keywords: Pneumology; idiopathic pulmonary fibrosis; progressive disease; combined therapy; pirfenidone; nintedanib
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Disease Progression | interventions — pirfenidone; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined therapy (Experimental)
  Interventions: Drug: pirfenidone and nintedanib
- Switch monotherapy (Active Comparator)
  Interventions: Drug: pirfenidone or nintedanib
- Control group (Other)
  Interventions: Drug: pirfenidone or nintedanib

INTERVENTIONS:
Drug: pirfenidone and nintedanib — The experimental group will receive pirfenidone 2403 mg per day (at least 1602 mg) in combination with nintedanib 300 mg per day (at least 200 mg) during 24 weeks.
  Arms: Combined therapy
Drug: pirfenidone or nintedanib — The second intervention group will switch from one monotherapy during 24 weeks: with pirfenidone 2403 mg per day (at least 1602 mg) or nintedanib 300 mg per day (at least 200 mg) to the other monotherapy (nintedanib in patients who received pirfenidone as first line therapy before inclusion and conversely).
  Arms: Switch monotherapy
Drug: pirfenidone or nintedanib — The control group will keep on the same monotherapy during 24 weeks: with pirfenidone 2403 mg per day (at least 1602 mg) or nintedanib 300 mg per day (at least 200 mg) to the other monotherapy (nintedanib in patients who received pirfenidone as first line therapy before inclusion and conversely).
  Arms: Control group

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a prototype of chronic, progressive, and fibrotic lung disease. It has been considered rare, with an incidence estimated to 11.5 cases per 100 000 individuals per year. Increasing rates of hospital admissions and deaths due to IPF suggest an increasing burden of disease. The median survival time from diagnosis is 2-4 years.

Recently two disease-modifying therapies, pirfenidone and nintedanib, have been approved worldwide. Both drugs reduce the disease progression as measured by progressive decline in forced vital capacity (FVC), with a reduction of overall mortality showed by meta-analysis of phase III pirfenidone trials.

However, progression of disease continues to occur despite the currently available drug therapy. Many patients die from progressive, chronic hypoxemic respiratory failure, or less frequently from acute exacerbation of pulmonary fibrosis. In these patients, no data are available to guide management between continuation of the prescribed antifibrotic drug, to switch to the other available antifibrotic drug, or to combine the available drugs.

The combination of nintedanib and pirfenidone is not recommended outside clinical trials. However, although both antifibrotic drugs were developed and approved as monotherapy, two recent trials have suggested the feasibility and safety of combining them over a 12-24 weeks period. These results encourage further studies of combination treatment with pirfenidone and nintedanib in patients with IPF. Such study is timely, as there is a risk that clinicians facing the continued worsening of disease in patients receiving one of the available drugs may prescribe both drugs combined outside clinical trials, potentially exposing patients to a currently unknown risk.

This study will evaluate the efficacy and tolerance of the combination pirfenidone and nintedanib as compared to a "switch monotherapy": i.e. switching from the current to the other of the two existing drugs prescribed as monotherapy, in patients who present chronic worsening IPF despite receiving either pirfenidone or nintedanib and as to a "control group": i.e.treatment still be on as before randomization (pirfenidone or nintedanib).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 50 years.
* Patient with Idiopathic Pulmonary Fibrosis satisfying the ATS/ERS/JRS/ALAT diagnostic criteria (29) diagnosed.

In the absence of a surgical lung biopsy, high-resolution computed tomography (HRCT) must be "consistent with Usual Interstitial Pneumonia (UIP)" defined as meeting either criteria A, B, and C, or criteria A and C, or criteria B and C below:

A. Definite honeycomb lung destruction with basal and peripheral predominance. B. Presence of reticular abnormality and traction bronchiectasis consistent with fibrosis, with basal and peripheral predominance.

C. Atypical features are absent, specifically nodules and consolidation. Ground glass opacity, if present, is less extensive than reticular opacity pattern.

* - Patient who fulfill at least 1 of the 4 criteria for IPF progression in the 12 months (+/- one six months) before screening, despite antifibrotic treatment in clinical practice (if yes check the option(s)). These criteria are: 0 Relative decline in FVC ≥10% predicted 0 Relative decline in FVC ≥5-<10% predicted and worsened respiratory symptoms 0 Relative decline in FVC ≥5-<10% predicted and increased extent of fibrotic changes on chest imaging 0 Worsened respiratory symptoms and increased extent of fibrotic changes on chest imaging
* Patient must have been on a stable dose of pirfenidone or nintedanib prescribed as first-line therapy for at least 6 months, with good tolerance of 1602 to 2403 mg per day of pirfenidone or 200 to 300 mg per day of nintedanib.
* Patient who has a FVC ≥ 45% of predicted.
* Patient who has a forced expiratory volume in 1 second (FEV1)/FVC ratio > 0.70.
* Patient who has a life expectancy of at least 9 months.
* Patient who has provided his written informed consent to participate in the study.
* Patient affiliated to a social insurance regimen.

Exclusion Criteria:

* Patients under judicial protection.
* Female patient who is pregnant or lactating, or is of child bearing potential (defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if ≤ 55 years or 12 months if > 55 years) and who did not agree to use highly effective methods of birth control throughout the study.
* Patient who is currently on both pirfenidone and nintedanib.
* Patient who has already received pirfenidone and nintedanib either concomitantly or successively.
* Patient who has a contra-indication to pirfenidone or nintedanib.
* Patient who has emphysema > 15% on HRCT or the extent of emphysema is greater than the extent of fibrosis according to reported results from the most recent HRCT.
* Patient who had acute exacerbation of idiopathic pulmonary fibrosis within the previous 3 months.
* Patient who has a history of cigarette smoking within the previous 3 months.
* Patient who has received experimental therapy for IPF within 4 weeks before baseline.
* Patient who is receiving systemic corticosteroids equivalent to prednisone > 15 mg/day or equivalent within 2 weeks before baseline.
* Patient who received Immuno-suppressants (e.g. methotrexate, azathioprine, cyclophosphamide, cyclosporine, sirolimus, everolimus or other immunosuppressants) within 4 weeks before baseline.
* Patient who has a history of a malignancy within the previous 5 years, with the exception of basal cell skin neoplasms. In addition, a malignant diagnosis or condition first occurring prior to 5 years must be considered cured, inactive, and not under current treatment.
* Patient who, in the Investigator's opinion, is not able to perform home spirometry in accordance with the protocol.
* Patient who has any concurrent condition other than IPF that, in the Investigator's opinion, is unstable and/or would impact the likelihood of survival for the study duration or the subject's ability to complete the study as designed, or may influence any of the safety or efficacy assessments included in the study.
* Patient who has baseline resting oxygen saturation of < 88% on room air or supplemental oxygen.
* Patient who had lung transplantation or who is on a lung transplant list and the investigator anticipates the patient will not be able to complete the study prior to transplant.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Slope of the decline in the forced vital capacity (FVC) measured by spirometry | 24 weeks
  FVC will be measured by spirometry

SECONDARY OUTCOMES:
The proportion of patients who continue intent-to-treat therapy | 24 weeks
  Tolerance of antifibrotic therapy at week 24, at a minimal daily dose of two thirds of the full treatment dose (e.g. 200 mg/day of nintedanib and/or 1602 mg/day of pirfenidone), with temporary interruptions of no more than 28 consecutive days.
Time to permanent study drug discontinuation | 24 weeks
  The interval from study treatment randomization to study drug permanent discontinuation or the end of follow-up. Study drug discontinuation will be considered in case of permanent termination of drug treatment allocated by randomization, transient discontinuation for longer than 28 consecutive days, or dose reduction below two thirds of the full treatment dose (i.e. 200 mg per day of nintedanib or 1602 mg per day or pirfenidone).
Time to treatment failure | 24 weeks
  The time from study treatment randomization to the first occurrence during the 24 weeks follow-up of any of the following events:
  * Death from any cause,
  * Non-elective hospitalization from pulmonary cause (which is predefined by a set of criteria in protocol),
  * Acute exacerbation of idiopathic pulmonary fibrosis (idiopathic or triggered),
  * Decrease (based on relative decline) from baseline of ≥ 10% in FVC,
  * Permanent study drug discontinuation (see above) (allcause). or the end of follow-up.
Proportion of decrease ≥ 10% FVC relative decline or death | 24 weeks
  Proportion of patients with ≥ 10% FVC relative decline or death at week 24.
Hospitalization-free survival | 24 weeks
  The time from randomization to the first occurrence during the 24 weeks follow-up of any of the following events:
  * Death from any cause,
  * All-cause unscheduled hospital admission, or the end of follow-up.
Time from randomization to the first non-elective hospitalization from pulmonary cause | 24 weeks
  Non-elective hospitalization from pulmonary cause (which is predefined by a set of criteria in protocol) during the 24 weeks follow-up or the end of follow-up.
Time from randomization to death | 24 weeks
  Time from randomization to death from any cause during the 24 weeks of the study or the end of follow-up.
Progression of disease on imaging by computed tomography | 24 weeks
  Progression of disease evaluated by the change from baseline in volume of fibrotic features at imaging by computed tomography assessed at 24 weeks.
Time from randomization to initiation of supplementary oxygen therapy | 24 weeks
  Time from randomization to initiation of supplementary oxygen therapy during the 24 weeks of the study or the end of follow-up.
Time from randomization to acute exacerbation of idiopathic pulmonary fibrosis | 24 weeks
  Time from randomization to acute exacerbation of idiopathic pulmonary fibrosis (idiopathic or triggered) during the 24 weeks of the study or the end of follow-up.
Quality of live assessed by the "Analogy and Likert" scale for the evaluation of dyspnea, cough and respiratory health | 24 weeks
  Absolute change in the "Analogy and Likert" scale relative to symptoms and impact on quality of life between baseline and week 24. The scale is between 3 and 11 points : 3 being the worst score and 11 being the best
Quality of live assessed by the "Pulmonary Fibrosis (L-PF)" questionnaire | 24 weeks
  Absolute change in Living with the "Pulmonary Fibrosis (L-PF)" questionnaire relative to symptoms and impact on quality of life between baseline and week 24.
Quality of live assessed by EuroQoL 5-dimension 5-level Questionnaire | 24 weeks
  Absolute change in EuroQoL 5-dimension 5-level (EQ-5D-5L) Questionnaire relative to symptoms and impact on quality of life between baseline and week 24. This questionnaire gives a score between 0 and 100 : 0 being the worst condition possible and 100 being the best.
Quality of live assessed by King's Brief Interstitial Lung Disease Questionnaire | 24 weeks
  Absolute change in King's Brief Interstitial Lung Disease Questionnaire (K-BILD) relative to symptoms and impact on quality of life between baseline and week 24. This questionnaire gives a score between 0 and 100 : 0 being the worst score and 100 being the best
Link between CA-125 variations and disease progression, the endpoint will be the slope of the FVC (exploratory) | 24 weeks
  For the analysis of the link between CA-125 variations and disease progression, the endpoint will be the slope of the FVC measured during 24 weeks by hospital spirometry. The CA-125 variations between baseline and 12 weeks will be categorized in two categories: increased versus stable or decreased.
Link between biomarkers variations and disease progression, the endpoint will be the slope of the FVC (exploratory) | 24 weeks
  For the analysis of the link between biomarkers variations and disease progression, the endpoint will be the slope of the FVC measured during 24 weeks by hospital spirometry. The biomarkers variations between baseline and 12 weeks will be categorized in two categories: increased versus stable or decreased. (Ancillary study)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent COTTIN, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (22):
- France (22):
  - CHU d'Angers, Angers
  - Centre Hospitalier de la côte Basque, Bayonne
  - CHRU de Besançon - Hôpital Jean Minjoz, Besançon
  - AP - HP - Hôpital Avicenne, Bobigny
  - CHRU Hôpital Cavale Blanche, Brest
  - Hôpital Pneumologique et Cardiovasculaire Louis Pradel, Bron
  - CHU de Caen - Hôpital de la Côte de Nacre, Caen
  - CHU Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - CHRU de Lille - Hôpital Albert Calmette, Lille
  - CHU de Marseille - Hôpital Nord, Marseille
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU - Hôpital G.R. Laennec, Nantes
  - CHU de Nice, Hôpital Pasteur, Nice
  - APHP - Hôpital Xavier Bichat-Claude Bernard, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - CHU Poitiers, Poitiers
  - Ch de Cornouaille, Quimper
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - CHRU, Tours - Hôpital Bretonneau, Tours
  - CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy
  - Hôpital Robert Schuman, Vantoux

IPD SHARING:
Plan to Share IPD: Undecided